CLINICAL TRIAL: NCT04997070
Title: Evaluation of Embryo Quality After Sperm Selection Using Microfluidic Technology: Study on Sibling Oocytes
Brief Title: Sperm Selection Using Microfluidic Technology
Acronym: MSS
Status: Completed | Type: Observational
Sponsor: CRG UZ Brussel (Other)
Responsible Party: Principal Investigator, Koen Wouters, Clinical Embryologist, CRG UZ Brussel
Other Study IDs: 2021-185
Record Dates: First submitted 2021-08-04; First posted 2021-08-09 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This clinical study has been organised to investigate whether microfluidic technology may be considered as a new procedure for routine sperm preparation during assisted reproduction. This is a technique that is already used in other centres.

The Microfluidic Sperm Sorting (MSS) technology reduces the time of sample preparation while selects a sperm population with better motility and less DNA fragmentation as compared to routine procedures. This med-ical device is already CE marked.

Having the intention to implement this technology in our department, we conduct this study to investigate whether the use of MSS has at least the same impact, if not better, on fertilization and embryo quality as compared to standard sperm selection procedures.

DETAILED DESCRIPTION:
To perform ICSI, the best spermatozoa are selected based on their motility. This is done using a standard procedure which is time-consuming and involves centrifugation steps known to induce sperm DNA damage. Just before ICSI, the selection of the sperm cell that will be injected into the egg is based on morphological assessment (at 400x inverted phase contrast microscopy). However, the spermatozoa with DNA damage cannot be identified using microscopic procedures and therefore cannot be excluded for ICSI. It was reported that the sperm cells with DNA damage have a negative impact on embryo development and are correlated with increased miscarriage rate.

A more "close to nature" approach is now available due to the microfluidic sperm sorting (MSS) technology that is using FERTILE series devices (FERTILE and FERTILE PLUS, Koek EU, GmbH). The method is based on the principle of natural sperm selection in a passage through micro-barriers imitating natural environment of female reproductive system (fallopian tubes).

This chemical-free technology does not require any pretreatment of the semen sample, while the sorted sperm shows high motility and low levels of DNA damage. At the day of pick up, the husband provides the semen sample. The sample obtained will be divided in 2 fractions: one fraction will be subject to Microfluidic technology (fraction 1) and the other fraction will represent the control (conventionally prepared sperm; fraction 2).

This device was tested in our laboratory on diagnostic semen samples and proved to select the best sperm population when compared to the standard method.

Due to the encouraging results, we intend to apply microfluidic as the routine procedure for sperm preparation in our department. This procedure will increase the chance of using sperm cells without DNA damage during ICSI and therefore we expect better embryological outcome.

This clinical study has been organised to determine if the embryo quality on day 5 will be similar or better when using microfluidic technology compared to standard procedure.

At the moment of ICSI, half of the eggs of good quality (mature) will be inseminated with sperm from fraction 1 and the other half with sperm from fraction 2. The decision of which fraction will be used to inject the first half of the oocytes is random and is based on a list generated by the computer.

The retrieved oocytes will follow the normal lab procedure after injection: the embryos available on day 3 or day 5/6 that meet our criteria for transfer or cryopreservation will be used for transfer or cryopreservation, no matter from which fraction the sperm was used.

ELIGIBILITY:
Inclusion Criteria:

* ICSI cycles planned for embryo transfer or 'freeze all' procedure
* Day 5 or day 3/5 embryo culture
* Fresh semen samples with ≥ 1x106 sperm/ml (raw) and Motility of 30% Grade A+B
* At least 6 follicles of ≥14 mm at the day of hCG administration
* Minimum 6 mature oocytes after oocyte pick up

Exclusion Criteria:

* Cycles with frozen semen sample
* Cycles with testicular sample
* In vitro fertilization (IVF) cycles
* In vitro maturation cycles
* Managed Natural Cycles (MNC)
* Egg bank- Acceptors
* PGT cycles

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Couples undergoing ICSI procedure in CRG UZ Brussel will be included in the trial if they fulfil the inclusion criteria listed.
Sampling Method: Probability Sample
Enrollment: 1038 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Embryo quality | 2 years
  Compare the embryo quality (Gardner score - Scale blastocyst 1-6 where 6 is best; Inner cell mass A-D where A is best; Throphectoderm A-C where A is best) on day 5 between the two groups.

SECONDARY OUTCOMES:
Fertilization rate | 2 years
  Compare the fertilization rate (number of fertilized oocytes per number of injected oocytes) between the two groups.
Embryo morphokinetic parameters | 2 years
  Compare the embryo morphokinetic parameters from day 0 until day 6 recorded via embryoscope Plus (Vitrolife sa) between the two group.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Wouters, Msc, Principal Investigator — Brussels IVF
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No